CLINICAL TRIAL: NCT07042854
Title: Volume-Controlled vs Pressure-Regulated Volume Control Ventilation in Pediatric Anesthesia: an Electrical Impedance Tomography Based Study
Acronym: VC_PRVC_ped
Status: Completed | Type: Observational
Sponsor: Vittore Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, Anna Camporesi, Medical Coordinator for Pediatric Anesthesia, Vittore Buzzi Children's Hospital
Other Study IDs: 2023/ST/099
Record Dates: First submitted 2025-06-11; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Ventilation Homogeneity; Anesthesia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single cohort: Each patient has received both ventilatory modes with same settings (tidal volume- TV, respiratory rate- RR, positive end expiratory pressure- PEEP- and inspired fraction of Oxygen - FiO2). Intra-lung compliance and global inhomogeneity Index (GI) were assessed though Electric Impedance Tomography (EIT) (PulmoVista 500, Draeger Medical, Germany), allowing at least five minutes after change of mode to let adequate time for gas distribution. At the same time, respiratory mechanics measures were obtained in quasi-static conditions after an inspiratory hold manoeuver, ensuring stability of plateau pressure (PPLAT). We assessed resistive (PIP-PPLAT) and elastic components (DeltaP and quasi-static compliance) of working pressure, and mechanical power as a marker of energy dissipation.

SUMMARY:
The primary goal of this prospective, observational crossover study is to investigate mechanical and EIT (Electrical Impedance Tomography) differences between Volume-Controlled Ventilation (VCV) and Pressure-Regulated Volume Controlled Ventilation (PRVC) in pediatric patients undergoing general anesthesia with endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists' status 1 and 2
* Provision of general anesthesia requiring endotracheal intubation

Exclusion Criteria:

* chronic lung diseases
* thoracic surgery
* thoracic or airway malformation
* presence of tracheostomy
* acute pulmonary conditions (secretions, laryngospasm, bronchoconstriction, pneumothorax) during anesthesia

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Healthy pediatric patients undergoing general anesthesia requiring endotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Intra-lung Compliance | Perioperatory.
  Intra-lung Compliance is an EIT- based parameter which shows if, between the two modes of ventilation, there is a net gain or loss of intraprenchimal compliance. This is expressed as percentage change from the first-point Compliance measured. We will compare Compliance in PRVC to RVD in VCV ventilation. VCV is the reference point.

SECONDARY OUTCOMES:
Global Inhmogeneity Index (GI) | Perioperatory.
  GI is a EIT-derived index to quantify the tidal volume distribution within the lung. We will compare GI in PRVC to RVD in VCV ventilation. VCV is the reference point.
Regional Ventilation Delay (RVD) | Perioperatory.
  RVD is an index of inhomogeneous ventilation. RVD quantifies the time difference between the onset of ventilation in different lung regions relative to a reference point. We will compare RVD in PRVC to RVD in VCV ventilation. VCV is the reference point.

CONTACTS AND LOCATIONS:
Locations (1):
- Vittore Buzzi Children's Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim YS, Won YJ, Lee DK, Lim BG, Kim H, Lee IO, Yun JH, Kong MH. Lung ultrasound score-based perioperative assessment of pressure-controlled ventilation-volume guaranteed or volume-controlled ventilation in geriatrics: a prospective randomized controlled trial. Clin Interv Aging. 2019 Jul 18;14:1319-1329. doi: 10.2147/CIA.S212334. eCollection 2019. PMID 31409981
- [Result] Camporesi A, Roveri G, Vetrugno L, Buonsenso D, De Giorgis V, Costanzo S, Pierucci UM, Pelizzo G. Lung ultrasound assessment of atelectasis following different anesthesia induction techniques in pediatric patients: a propensity score-matched, observational study. J Anesth Analg Crit Care. 2024 Oct 5;4(1):69. doi: 10.1186/s44158-024-00206-x. PMID 39369249
- [Result] Wang Q, Li Y, Zhao K, Zhang J, Zhou J. Optimizing perioperative lung protection strategies for reducing postoperative respiratory complications in pediatric patients: a narrative review. Transl Pediatr. 2024 Nov 30;13(11):2043-2058. doi: 10.21037/tp-24-453. Epub 2024 Nov 26. PMID 39649647
- [Result] Nascimento MS, Rebello CM, Costa ELV, Correa LC, Alcala GC, Rossi FS, Morais CCA, Laurenti E, Camara MC, Iasi M, Apezzato MLP, do Prado C, Amato MBP. Effect of general anesthesia and controlled mechanical ventilation on pulmonary ventilation distribution assessed by electrical impedance tomography in healthy children. PLoS One. 2023 Mar 16;18(3):e0283039. doi: 10.1371/journal.pone.0283039. eCollection 2023. PMID 36928465